CLINICAL TRIAL: NCT00586170
Title: A Prospective, Randomized, Double-Blind Study on Adjunctive Use of Pulsed Electromagnetic Fields in the Treatment of 5th Metatarsal Non-Union Fractures: Effect on Clinical Outcome and Growth Factor Synthesis
Brief Title: A Double-Blind Study on Adjunctive Use of PEMF in the Treatment of 5th Metatarsal Non-Union Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-027
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Nonunion of Fracture of Fifth Metatarsal
Keywords: nonunion; fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBI Bone Healing System + Surgery (Experimental): Subject will be using the EBI Bone Healing System (active device) in conjunction with ORIF surgery of the nonunion site.
  Interventions: Device: EBI Bone Healing System; Procedure: Surgery
- Placebo Device + Surgery (Placebo Comparator): Subject will be using a placebo device in conjunction with ORIF surgery of the nonunion site.
  Interventions: Device: Placebo Device; Procedure: Surgery

INTERVENTIONS:
Device: EBI Bone Healing System — 10 hours of treatment per day for up to 24 weeks
  Arms: EBI Bone Healing System + Surgery
Device: Placebo Device — 10 hours of treatment per day for up to 24 weeks
  Arms: Placebo Device + Surgery
Procedure: Surgery — Open Reduction and Internal Fixation of the nonunion site

SUMMARY:
The purpose of this study is to analyze the effect of PEMF in surgical reconstruction of 5th metatarsal non-union fractures.

DETAILED DESCRIPTION:
The investigators hypothesize:

1. That treatment of 5th metatarsal non-union fracture with PEMF will achieve earlier resolution and/or higher success compared to surgery alone of 5th metatarsal non-union fractures.
2. PEMF will stimulate increased expression of critical growth factors (i.e. BMP-2, BMP-4, BMP-7 as well as TGFb, IGF-1, FGF-2 and VEGF) at the non-union site to facilitate osseous healing of 5th metatarsal non-union fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been diagnosed with a 5th metatarsal delayed or non-union.
2. Subjects with duration of a 5th metatarsal fracture for a minimum of 3 months.
3. Male or female between ages of 18 and 75 years old, inclusive

Exclusion Criteria:

1. Subject has synovial pseudarthrosis.
2. Subject has a fracture gap of larger than 5mm as measured on CT Scan.
3. Subjects with conditions associated with elevated circulatory levels of inflammatory cytokines e.g., multiple trauma.
4. If female, subject is pregnant, plans on becoming pregnant during the duration of this clinical outcomes collection study or lactating.
5. Subject has an implanted unipolar pacemaker.
6. Subjects who have previous malignant or connective tissue disorder.
7. Subjects who use medication such as steroids or anticoagulants.
8. Subjects who have an underlying osseous infection (Osteomyelitis) and/or open wound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-11; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Evangelista, Study Director — Zimmer Biomet
Locations (2):
- United States (2):
  - Neurological Institute of NJ, Newark, New Jersey
  - The Orthopedic Foot and Ankle Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EBI Bone Healing System + Surgery | Placebo Device + Surgery
Started | 5 | 3 (Initially enrollment was listed as 9. 1 placebo patient withdrew prior to surgery, so enrollment=8.)
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EBI Bone Healing System + Surgery | Placebo Device + Surgery | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful 5th Metatarsal Unions Achieved.
Description: Each patient was assessed radiographically at 2, 4, 6, 8, 12, 16, 20, and 24 weeks or until radiographic signs of healing were evident. The radiographs were evaluated and graded by the number of cortices (medial and lateral on anteroposterior views as well as dorsal and plantar on lateral views) of healing at each time point. Bridging callus across 4 cortices on postoperative radiographs was used to determine healing.
Time Frame: 24 Weeks
Population: Each patient had 1 fracture. The number of fractures treated equals the number of patients treated in both treatment groups.
Measure: Number; unit: percentage of fractures healed
Units Other Than Participants: Fractures
Arm/Group | EBI Bone Healing System + Surgery | Placebo Device + Surgery
Number analyzed (Participants) | 5 | 3
Number analyzed (Fractures) | 5 | 3
percentage of fractures healed | 100 | 100

2. Secondary Outcome: Mean AOFAS Score (% Change From Baseline), Foot Function Index (% Change From Baseline), SF-36 Health Survey (Change From Baseline)
Time Frame: 24 Weeks
Population: No AOFAS, Foot Function Index, or SF-36 Health Survey data was collected or analyzed.
Arm/Group | EBI Bone Healing System + Surgery | Placebo Device + Surgery
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Entire study period. Patients were followed through healing, or up to 24 weeks.
Arm/Group | EBI Bone Healing System + Surgery | Placebo Device + Surgery
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 3/5 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBI Bone Healing System + Surgery (N=5) | Placebo Device + Surgery (N=3)
Unrelated complication - leg bruising, breast lump (Investigations) | 0 (0) | 1 (1) — 2 months post surgery patient had a lump in left breast and severe bruising on right leg. Could not be associated with device use.
Unrelated complication - anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — increased anxiety due to cast reported 3 weeks post-surgery. Patient recovered.
unrelated complication - hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) — patient had vomiting and hernia obstruction 6 weeks post-surgery; had hernia surgery and recovered
unrelated complication - allergic reaction (General disorders) | 1 (1) | 0 (0) — patient had sick stomach on surgery day, 3 days later reported allergic reaction - increased swelling of the face, hands and legs. Discontinued medication and swelling discontinued. Vomiting and diarrhea reported 3 wks post-surgery. patient recovered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No